CLINICAL TRIAL: NCT06804889
Title: Effect of Cannabidiol-Based Vaginal Suppositories on Menopausal Symptoms: a Randomized Double-Blind Placebo-Controlled Clinical Trial Using MRS and MANSA Questionnaires
Brief Title: Effect of CBD-Based Vaginal Suppositories on Menopausal Symptoms
Acronym: Gyno-CBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Collaborators: CB21 Pharma Ltd. (Unknown)
Responsible Party: Principal Investigator, Jan Vacek, Olomouc University Hospital, Palacky University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 194/22
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Menopause and Genitourinary Syndrome
Keywords: menopause, quality of life, cannabidiol, hyaluronic acid, vaginal suppositories

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Received placebo vaginal suppositories.
  Interventions: Device: Placebo Suppositories
- CANNEFF® VAG SUP (Active Comparator): Received CANNEFF® VAG SUP vaginal suppositories.
  Interventions: Device: CANNEFF® VAG SUP vaginal suppositories

INTERVENTIONS:
Device: CANNEFF® VAG SUP vaginal suppositories — CANNEFF® VAG SUP vaginal suppositories containing 100 mg cannabidiol - CBD and 6.6 mg hyaluronic acid - HA.
  Arms: CANNEFF® VAG SUP
Device: Placebo Suppositories — Received placebo vaginal suppositories with identical composition as for Active Comparator, but without both active ingredients (CBD - cannabidiol and HA - hyaluronic acid).
  Arms: Placebo

SUMMARY:
Efficacy and safety of the medical device CANNEFF® vaginal suppositories containing two active ingredients cannabidiol (CBD) and hyaluronic acid (HA) in alleviating menopausal symptoms and improving quality of life in (post)menopausal women will be evaluated.

DETAILED DESCRIPTION:
Current state of the art: Menopause is a significant transitional phase in a woman's life, marked by the cessation of ovarian function and a decline in estrogen levels, typically occurring between the ages of 40 and 55. This hormonal shift leads to various physiological and psychological symptoms, including hot flashes, sleep disturbances, mood swings, anxiety, depression, fatigue, and sexual dysfunction. These symptoms can profoundly impact daily activities and interpersonal relationships.

Study description: The study was designed as a randomised, double-blind, placebo-controlled clinical trial conducted at the Gynaecology and Obstetrics Clinic Meda, Prague 8, Czech Republic. The study adhered to the Consolidated Standards of Reporting Trials (CONSORT) guidelines and the principles of the Declaration of Helsinki (1975, revised in 2013). Baseline assessments included MRS, MANSA questionnaires, hormone levels (FSH, LH, estradiol), and the CA-125. These assessments were repeated at the end of the 30-day treatment period for the MRS, MANSA scores, and CA-125 analysis. The primary outcome measures were the changes in MRS and MANSA scores from baseline to post-treatment. Secondary outcomes included changes in the CA-125 marker, as well as any adverse events reported during the study period.

Recruitment and study: Post/menopausal women presenting with significant climacteric symptoms and reporting partner sexual discomfort were initially assessed. Inclusion criteria included women older than 40y experiencing (post)menopausal symptoms and absence of microbial infection. Exclusion criteria included a history of gynaecological oncology, diabetes, current treatment with antidepressants, antibiotics, or any contraindications to vaginal suppository use, as well as users of cannabis or cannabis products.

Intervention: Participants were randomized into two groups: Group A received CANNEFF® vaginal suppositories containing 100 mg CBD and 6.6 mg HA per one suppository, and Group B received placebo suppositories of identical composition without the active ingredients. Both groups used one suppository for nightly for 30 days.

Evaluation of study results: Pre-treatment and post-treatment assessments included the Menopause Rating Scale (MRS) and the Manchester Short Assessment of Quality of Life (MANSA) validated questionnaires and the CA-125 marker monitoring. Hormone levels (FSH, LH, estradiol) were measured during pre-treatment assessments to confirm menopausal status. Secondary outcomes included changes in the CA-125 marker and any adverse events reported during the study.

ELIGIBILITY:
Inclusion Criteria:

Women experiencing (post)menopausal symptoms and absence of microbial infection.

Exclusion Criteria:

Women with history of gynaecological oncology, diabetes, current treatment with antidepressants, antibiotics, or any contraindications to vaginal suppository use, as well as users of cannabis or cannabis products.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological female identity.
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Alleviating menopausal symptoms in (post)menopausal women | 12 months
  The primary outcome measure was the changes in MRS (Menopause Rating Scale) scores from baseline to post-treatment. The MRS questionnaire covers 11 symptoms in somatic-vegetative, psychological and urogenital domains. The respondents evaluate the intensity of the various symptoms using a Likert scale 0-4 (0 - none; 1 - minor; 2 - medium; 3 - major; 4 - unbearable difficulties).
Improving quality of life in (post)menopausal women | 12 months
  The primary outcome measure was the changes in MANSA (Manchester Short Assessment of Quality of Life) scores from baseline to post-treatment. 16-item questionnaire evaluating quality of life was used, rated from 1 (could not be worse) to 7 (could not be better).

SECONDARY OUTCOMES:
Safety profile evaluation via adverse events reported | 12 months
  The secondary outcome measure was the number of adverse events reported during the study period by patients or physician.
Safety profile evaluation via CA-125 pathology marker analysis | 12 months
  The secondary outcome measure was the changes in CA-125 marker monitored. CA-125 is a pathology marker commonly used in gynecology, with a reference range of 0 to 35 kU/L. Within this range = no pathology during the intervention. The value > 35 kU/L = pathological changes during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynaecology and Obstetrics Clinic Meda, Prague, Czechia, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Priebe S, Huxley P, Knight S, Evans S. Application and results of the Manchester Short Assessment of Quality of Life (MANSA). Int J Soc Psychiatry. 1999 Spring;45(1):7-12. doi: 10.1177/002076409904500102. PMID 10443245
- [Background] Pisanti S, Malfitano AM, Ciaglia E, Lamberti A, Ranieri R, Cuomo G, Abate M, Faggiana G, Proto MC, Fiore D, Laezza C, Bifulco M. Cannabidiol: State of the art and new challenges for therapeutic applications. Pharmacol Ther. 2017 Jul;175:133-150. doi: 10.1016/j.pharmthera.2017.02.041. Epub 2017 Feb 22. PMID 28232276
- [Background] Marino JL, Saunders CM, Emery LI, Green H, Doherty DA, Hickey M. Nature and severity of menopausal symptoms and their impact on quality of life and sexual function in cancer survivors compared with women without a cancer history. Menopause. 2014 Mar;21(3):267-74. doi: 10.1097/GME.0b013e3182976f46. PMID 23860358